CLINICAL TRIAL: NCT04273802
Title: CPX-351 in Higher Risk Myelodysplastic Syndromes: a Phase I/ II Study as First Line or After Hypomethylating-agents Failure
Brief Title: CPX-351 in Higher Risk Myelodysplastic Syndromes
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Groupe Francophone des Myelodysplasies (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GFM-CPX-MDS
Record Dates: First submitted 2020-02-12; First posted 2020-02-18 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Myelodysplastic Syndromes
Keywords: MDS high risk
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — CPX-351

STUDY DESIGN:
Intervention Model Description: Cohort A: first line treatment Cohort B: after hypomethylating-agents failure
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A - First line treatment (Experimental): Untreated patients
  Interventions: Drug: CPX-351 in cohort A
- Cohort B - Hypomethylating failure (Experimental): Patients in absence of response after hypomethylating agents treatment
  Interventions: Drug: CPX-351 in cohort B

INTERVENTIONS:
Drug: CPX-351 in cohort A — Treatment by CPX-351 via intravenous infusion over 90 minutes.
  Induction treatment with CPX-351 100 Units/m²/D on days 1, 3 and 5.
  If response after this induction treatment, 4 courses of consolidation therapy with CPX-351 100 Units/m²/D on day 1.
  If no response after this induction treatment, a second induction course of CPX-351 100 Units/m²/D on days 1 and 3. If response is achieved after this salvage course, 3 courses of consolidation therapy with CPX-351 100 Units/m²/D on day1.
  Arms: Cohort A - First line treatment
Drug: CPX-351 in cohort B — Treatment by CPX-351 via intravenous infusion over 90 minutes.
  This will be a dose-finding study : CPX-351 100 Units/m²/D on days 1, 3 and 5 or CPX-351 100 Units/m²/D on days 1 and 3 or CPX-351 60 Units/m²/D on days 1 and 3.
  In response after induction treatment, 4 monthly courses of consolidation therapy with CPX-351 at the same dose on day 1.
  Arms: Cohort B - Hypomethylating failure

SUMMARY:
Study of the efficacy of CPX-351 treatment in patients with higher risk myelodysplastic syndromes : as first line treatment or after hypomethylating agents failure

DETAILED DESCRIPTION:
A phase I/II study of the efficacy of CPX-351 treatment in patients with higher risk myelodysplastic syndromes : as first line treatment or after hypomethylating agents failure.

CPX-351 is an advanced liposomal formulation of daunorubicin and cytarabine encapsulated at a 1:5 ratio.

Patients will receive induction treatment with CPX-351. Patients in response (complete response (CR), complete response with incomplete hematologic improvement (CRi), partial response (PR)) after induction will receive monthly courses of consolidation therapy with CPX-351.

ELIGIBILITY:
Inclusion Criteria:

* Myelodysplastic syndrome (WHO 2016 classified) including CMML (even if white blood cell count (WBC) > 13000/mm3).
* For COHORT A: untreated patients except by erythropoiesis stimulating agents, Lenalidomide or non-chemotherapy during a phase of lower risk MDS; For COHORT B: absence of response (CR, CRi, PR or HI according to international working group (IWG) 2006 for MDS) after a minimum of 6 cycles of single hypomethylating agent or relapse after a response.
* For COHORT A: less than 20% of marrow blasts. For COHORT B: less than doubling of marrow blasts compared with onset of hypomethylating agent.
* Classical international prognostic scoring system (IPSS) int-2 or high risk score.
* For COHORT A and B : age between 18 and 70 years
* For COHORT A: Performance status (ECOG grading) ≤ 1; For COHORT B: Performance status ≤ 2.
* Eligible for standard intensive chemotherapy.
* Absence of concomitant severe cardiovascular disease which would make intensive chemotherapy impossible, i.e. arrhythmias requiring chronic treatment, congestive heart failure or symptomatic ischemic heart disease, reduced left ventricular function assessed by multigated acquisition (MUGA) scan or echocardiogram.
* Patient must have adequate organ function as indicated by the following laboratory values: Renal: Serum creatinine < 2 mg/dl or calculated creatinine clearance ≥ 60 mL/min by MDRD (modification of the diet in renal disease) or CKD-EPI (chronic kidney disease epidemiology collaboration) equation for patients with creatinine levels > 1.5xULN ; Hepatic: Serum total bilirubin ≤ 2.5xULN OR direct bilirubin ≤ ULN for patients with total bilirubin levels ≥ 2 mg/dL, aspartate aminotransferase (ALT) and alanine aminotransferase (ALT) ≤ 2.5xULN, Alkaline Phosphatase ≤ 5xULN (if > 2.5xULN, then liver fraction should be ≤ 2.5xULN).
* Patients not known to be refractory to platelet transfusions.
* Female subjects of child-bearing potential must agree to undergo medically supervised pregnancy test prior to starting study drug. The first pregnancy test will be performed at screening (within 7 days prior to first study drug administration), and on the day of the first study drug administration and confirmed negative prior to dosing and Day 1 before dosing all subsequent cycles. Female patient is not actively breastfeeding at the time of study entry.
* Female patients are either post-menopausal, free from menses for > 2 years, surgically sterilized or willing to use 2 adequate barrier methods of contraception to prevent pregnancy or agree to abstain from becoming pregnant throughout the study, starting with Visit 1. Females of reproductive potential as well as fertile men and their partners who are female of reproductive potential must agree to abstain from sexual intercourse or to use two highly effective forms of contraception from the time of giving informed consent, during the study and for 6 months (females and males) following the last dose of CPX-351.
* Male patients agree to use an adequate method of contraception for the duration of the study. Men should be advised not to father a child while receiving CPX-351 and for 6 months post study.
* Patients are available for regular blood sampling, study related assessments, and appropriate clinical management at the treating institution for the duration of the study.
* Patients have the ability to understand and willingness to sign an informed consent form indicating the investigational nature of the study.

Exclusion Criteria:

* Active and uncontrolled infection.
* Last dose of hypomethylating agent given more than 4 months before entering the trial.
* Uncontrolled intercurrent illness or circumstances that could limit compliance with the study, including but not limited to the following: symptomatic congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmia, pancreatitis, or psychiatric or social conditions that may interfere with patient compliance.
* Current participation or participation in a study with an investigational compound or device within 30 days of initial dosing with study drug.
* Known human immunodeficiency virus (HIV) infection or HIV-related malignancy.
* Clinically active hepatitis B or hepatitis C infection.
* Known allergy or hypersensitivity to any component of CPX-351.
* "Currently active" second malignancy, other than non-melanoma skin cancer and in situ carcinoma of the cervix.
* Subjects with a history of Wilson's disease or other copper-related disorder.
* Treatment with growth factors such as erythropoietin alfa (EPO) or granulocyte colony-stimulating factor (G-CSF) or cytotoxic and non-cytotoxic agents (including low dose oral chemotherapy with the exception of hydroxyurea) in the 30 days before inclusion.
* Treatment with systemic steroids that has not been stabilized to the equivalent of ≤ 10 mg/day prednisone during the 4 weeks prior to the start of the study drugs.
* Clinical evidence of central nervous system leukemia.
* Pregnancy or breastfeeding during the projected duration of the study.
* Absence of social security.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-04-29 (Actual); Primary Completion 2021-08-27 (Actual); Study Completion 2022-07-06 (Actual)

PRIMARY OUTCOMES:
Response rate (CR, CRi, PR) | 28 to 42 days after induction
  Response to induction therapy

SECONDARY OUTCOMES:
Overall response rate (CR, CRi, PR, HI) | 28 to 42 days after induction
  Response to induction therapy
Event free survival | 42 months
  Event free survival
Response duration | 42 months
  Duration of the response to induction therapy
Overall survival | 42 months
  Overall survival
Toxicity profile - Duration of cytopenias | 42 months
  Duration of cytopenias
Toxicity profile - life threatening or fatal cytopenias | 42 months
  Number of life threatening or fatal cytopenias
Toxicity profile - hospitalization | 42 months
  Time spent in hospital for induction and consolidation cycles
Evaluation of minimal residual disease (MRD) after induction and after the last consolidation | 42 months
  Evaluation of MRD by flow cytometry
Evaluation of minimal residual disease (MRD) after induction and after the last consolidation | 42 months
  Evaluation of variant allelic frequency (VAF) of Baseline mutations
Soluble Fms-like tyrosine kinase 3 ligand concentration (sFLc) in plasma during induction | 42 months
  sFLc plasma level assessments at day 1 of induction just before starting treatment, and then at days 8, 15 and 22 of induction

CONTACTS AND LOCATIONS:
Overall Officials: Pierre PETERLIN, MD, Principal Investigator — Nantes University Hospital
Locations (16):
- France (16):
  - CHU d'Amiens - Service d'hématologie clinique et thérapie cellulaire, Amiens
  - CHU d'Angers - Service des maladies du sang, Angers
  - Centre hospitalier Victor Dupouy - Service d'Hématologie, Argenteuil
  - CHU de Besançon - Hôpital Jean Minjoz - Service d'hématologie clinique, Besançon
  - CHU de Grenoble - Clinique universitaire d'hématologie, Grenoble
  - CH Le Mans - Service d'onco-hématologie, Le Mans
  - CHRU de Limoges - Hôpital Dupuytren - Service d'hématologie clinique et thérapie cellulaire, Limoges
  - Institut Paoli Calmettes - Unité d'hématologie 3, Marseille
  - CHU Hôtel Dieu - Service d'Hématologie Clinique, Nantes
  - CHU-Hôpital Archet I - Service d'Hématologie Clinique, Nice
  - Hôpital Saint Louis - Service Hématologie Séniors, Paris
  - CHU de Bordeaux - Hôpital de Haut-Lévêque - Service des maladies du sang, Pessac
  - CHU de Poitiers - Service d'onco-hématologie et thérapie cellulaire, Poitiers
  - Hôpital Pontchaillou - Service d'hématologie clinique, Rennes
  - Institut de Cancérologie Lucien Neuwirth - Hématologie Clinique - Thérapie Cellulaire, Saint-Priest-en-Jarez
  - IUCT-oncopole - Fédération Hématologie - Médecine Interne, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Peterlin P, Le Bris Y, Turlure P, Chevallier P, Menard A, Gourin MP, Dumas PY, Thepot S, Berceanu A, Park S, Hospital MA, Cluzeau T, Bouzy S, Torregrosa-Diaz JM, Drevon L, Sapena R, Chermat F, Ades L, Dimicoli-Salazar S, Chevret S, Bene MC, Fenaux P. CPX-351 in higher risk myelodysplastic syndrome and chronic myelomonocytic leukaemia: a multicentre, single-arm, phase 2 study. Lancet Haematol. 2023 Jul;10(7):e521-e529. doi: 10.1016/S2352-3026(23)00090-X. Epub 2023 May 25. PMID 37245522